CLINICAL TRIAL: NCT07327437
Title: Arthroscopic Trans-osseous Rotator-Cuff Repair Using the Giant-Needle and Grand-Knot Technique.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sherif Hamdy Zawam (Other)
Responsible Party: Sponsor-Investigator, Sherif Hamdy Zawam, Assistant Professor of Orthopedic Surgery, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB: 11625-442021
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Rotator Cuff Tear
Keywords: Rotator cuff; Transosseous; Giant needle; Grand Knot
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: This is a prospective, two-arm, parallel-group randomized comparative study. Participants were allocated to either the Experimental Group (arthroscopic trans-osseous repair using the 'Grand-Knot' suture-block technique) or the Active Comparator Group (arthroscopic repair using all-suture anchors) in a 1:1 ratio. Randomization was achieved via a computer-generated sequence. Allocation concealment was maintained using sequentially numbered, sealed opaque envelopes opened by an independent assistant only after the intraoperative confirmation of tear morphology. Both groups followed an identical, standardized postoperative rehabilitation protocol and were assessed at predetermined intervals up to 30 months.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grand-Knot Group (Experimental): Patients undergoing arthroscopic trans-osseous rotator cuff repair using the Grand-Knot suture-block technique.
  Interventions: Procedure: Grand-Knot Technique
- Suture Anchor Group (Active Comparator): Patients undergoing standard arthroscopic rotator cuff repair using all-suture anchors.
  Interventions: Device: All-Suture Anchors (Y-Knot RC)

INTERVENTIONS:
Procedure: Grand-Knot Technique — Use of a Giant-needle to create trans-osseous tunnels and securing the tendon with a specialized suture-block (Grand-Knot).
  Arms: Grand-Knot Group
Device: All-Suture Anchors (Y-Knot RC) — Standard repair using 2.8 mm all-suture anchors placed in the humeral footprint.
  Arms: Suture Anchor Group

SUMMARY:
The purpose of this study is to compare a novel, cost-effective arthroscopic trans-osseous rotator cuff repair technique, known as the 'Grand-Knot' technique, against the standard repair using all-suture anchors. The study evaluates which method provides better functional recovery and structural healing for patients with full-thickness supraspinatus tears. Patients were randomized to receive either the Grand-Knot repair or the standard anchor repair and were followed for a minimum of 2.5 years to assess shoulder function using the ASES score, range of motion, and tendon integrity."

DETAILED DESCRIPTION:
"This prospective randomized comparative study was designed to evaluate the clinical and biomechanical effectiveness of an anchorless trans-osseous repair for rotator cuff tears.

Participants: 160 patients (aged 45-75) with full-thickness supraspinatus or posterosuperior tears were enrolled.

Interventions: > 1. Experimental Group: The Grand-Knot technique utilized a 'Giant Needle' to create trans-osseous tunnels, through which sutures were passed and secured using a specialized suture-block (Grand-Knot) on the lateral cortex. 2. Control Group: Standard arthroscopic repair was performed using 2.8 mm all-suture anchors (Y-Knot RC).

Procedure: All surgeries were performed arthroscopically by a single senior surgeon. Postoperative rehabilitation was standardized for both groups.

Outcomes: The primary endpoint was the American Shoulder and Elbow Surgeons (ASES) score at 30 months. Secondary endpoints included the Constant score, objective range of motion (ROM) measured by a goniometer, and structural integrity of the tendon as assessed by postoperative MRI or ultrasound at 6 months. Additionally, the study incorporates biomechanical data comparing the load-to-failure strength of both constructs."

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 45 to 75 years.

Diagnosis of full-thickness supraspinatus or posterosuperior rotator-cuff tears.

Tears suitable for arthroscopic repair.

Confirmation of diagnosis and tear morphology via standardized clinical examination and MRI.

Willingness to comply with a 2.5-year follow-up protocol and standardized rehabilitation.

Exclusion Criteria:

* Partial-thickness tears or isolated subscapularis tears.

Advanced fatty infiltration (Fuchs grade 3-4).

Rotator cuff arthropathy (Hamada classification > 2).

Presence of calcific tendinitis in the affected shoulder.

Prior ipsilateral shoulder surgery.

General medical contraindications to arthroscopy or general anesthesia.

Inability to complete the follow-up or provide informed consent.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons ASES Score | 30 months (2.5 years) postoperatively
  The ASES score is a standardized clinician-completed and patient-reported instrument consisting of two sections: pain (50%) and activities of daily living (50%). The total score ranges from 0 to 100, where 100 indicates the best possible shoulder function and 0 indicates the worst.

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Zawam, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo University Hospitals (Kasr Al-Ainy), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share individual participant data has not yet been finalized. Access to de-identified data may be considered upon reasonable request to the Principal Investigator, subject to approval by the Cairo University Faculty of Medicine Research Ethics Committee and in accordance with institutional data privacy policies.

REFERENCES:
- [Background] Park MC, ElAttrache NS, Tibone JE, Ahmad CS, Jun BJ, Lee TQ. Part I: Footprint contact characteristics for a transosseous-equivalent rotator cuff repair technique compared with a double-row repair technique. J Shoulder Elbow Surg. 2007 Jul-Aug;16(4):461-8. doi: 10.1016/j.jse.2006.09.010. Epub 2007 Feb 22. PMID 17321161
- [Background] Richards RR, An KN, Bigliani LU, Friedman RJ, Gartsman GM, Gristina AG, Iannotti JP, Mow VC, Sidles JA, Zuckerman JD. A standardized method for the assessment of shoulder function. J Shoulder Elbow Surg. 1994 Nov;3(6):347-52. doi: 10.1016/S1058-2746(09)80019-0. Epub 2009 Feb 13. PMID 22958838
- [Background] Dines JS, et al. Biomechanical comparison of all-suture anchors and traditional rigid anchors. Arthroscopy. 2016.
- [Background] Author et al. Arthroscopic trans-osseous rotator cuff repair using the Grand-Knot technique: A technical note. Journal Name. Year.